CLINICAL TRIAL: NCT03570190
Title: Registry to Evaluate the Impact of a Valve Coordinator on Aortic Stenosis / TAVI Outcome - (German Pilot)
Acronym: Coordinate
Status: Completed | Type: Observational
Sponsor: Institut für Pharmakologie und Präventive Medizin (Network)
Collaborators: Edwards Lifesciences (Industry)
Responsible Party: Sponsor
Other Study IDs: Coordinate
Record Dates: First submitted 2018-03-23; First posted 2018-06-26 (Actual); Last update posted 2022-05-18 (Actual); Status verified 2022-05

CONDITIONS: Aortic Valve Stenosis
MeSH Terms: conditions — Aortic Valve Stenosis

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 30 Days
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- TAVI patients: elective patients with a diagnosis of sAS and admitted for TAVI attending one of the participating centers for commercially available balloon expandable valve implantation that will be managed by a coordinator
  Interventions: Other: Coordinator

INTERVENTIONS:
Other: Coordinator — A THV coordinator will be responsible for communication with the patients and the caregivers as well as for monitoring medical documentation and treatment pathways. The registry will consist of 3 phases:
  * Determination of the status quo
  * Dedicated reflection and training followed by implementation of tailored changes
  * Determination of the effect

SUMMARY:
Prospective, multicenter registry in patients undergoing commercially available balloon expandable valve implantation. The registry will consist of 3 phases:

Prospective determination of baseline Status Quo (3 months):

Documentation of treatment pathways and endpoints of "routine" patients without educational program

Dedicated reflection and training (1 day):

One training session after the observational period to reflect on treatment pathways, exchange between valve coordinators involved, and develop improvements.

Implementation of tailored changes (2 months):

Implementation of the changes developed in the training.

Determination of the effect (3 months):

Coordinator measures optimization changes and determines effects.

DETAILED DESCRIPTION:
Along the severe aortic stenosis (sAS) treatment pathway there are delays that may impact quality management and hospital efficiency. A dedicated valve coordinator, interfering with all stages of patient handling throughout the hospital may increase the efficiency of the sAS patient flow, accelerate decision making and clinical outcomes while at the same time decreasing resource consumption.

The hypothesis is that the implementation of a dedicated valve coordinator will improve the patient flow of sAS patients scheduled to undergo TAVI, their outcome, patient and physician satisfaction and will optimize costs.

In total, three centers across Germany (Munich, Düsseldorf, Bad Bevensen) will participate.

ELIGIBILITY:
Inclusion Criteria:

* elective patients with a diagnosis of severe symptomatic aortic stenosis and admitted for TAVI

Exclusion Criteria:

* patients not providing written informed consent

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Consecutive elective patients with a diagnosis of severe symptomatic aortic stenosis and admitted for TAVI attending one of the participating centers for commercially available balloon expandable valve implantation will be recruited.
Sampling Method: Non-Probability Sample
Enrollment: 161 (Actual)
Dates: Start 2018-12-20 (Actual); Primary Completion 2019-12-19 (Actual); Study Completion 2019-12-19 (Actual)

PRIMARY OUTCOMES:
Evaluation of differences in length of stay (LoS) | 12 months
  LoS in days.
Adverse event rate | 30 days
  According to VARC-2 criteria.
Patient satisfaction | 30 days
  Satisfaction score. The total score range is from 0 (extremely dissatisfied) to 40 (extremley satisfied).
Economic evaluation | 12 months
  Proportion of early discharges in patients with sAS undergoing TAVI.

CONTACTS AND LOCATIONS:
Overall Officials: Katja Bohmann, MD, Principal Investigator — Herz- u. Gefässzentrum Bad Bevensen
Locations (3):
- Germany (3):
  - Deutsches Herzzentrum München, München, Bavaria
  - Herz- u. Gefässzentrum Bad Bevensen, Bad Bevensen, Lower Saxony
  - Herz- und Gefäßzentrum, Düsseldorf, North Rhine-Westphalia

IPD SHARING:
Plan to Share IPD: No
no IPD will be shared

REFERENCES:
- [Result] Bohmann K, Burgdorf C, Zeus T, Joner M, Alvarez H, Berning KL, Schikowski M, Kasel AM, van Mark G, Deutsch C, Kurucova J, Thoenes M, Frank D, Wundram S, Bramlage P, Miller B, Veulemans V. The COORDINATE Pilot Study: Impact of a Transcatheter Aortic Valve Coordinator Program on Hospital and Patient Outcomes. J Clin Med. 2022 Feb 23;11(5):1205. doi: 10.3390/jcm11051205. PMID 35268296